CLINICAL TRIAL: NCT03288779
Title: Theta Burst Stimulation for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083070
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Theta Burst Stimulation Arm (Other): This is a pilot open label study.
  Interventions: Device: Theta Burst Stimulation

INTERVENTIONS:
Device: Theta Burst Stimulation — Transcranial magnetic stimulation with theta burst stimulation

SUMMARY:
Purpose and objective Schizophrenia is a chronic debilitating illness with cognitive deficits that cause serious impairment in psychosocial recovery and with few treatments to remediate these deficits. One area that holds great promise for the development of novel, effective therapies is noninvasive brain stimulation. The investigators have used one form of brain stimulation, transcranial magnetic stimulation (TMS), for some time to modulate and enhance cognitive function in the brain, especially working memory (WM) function, which has a central role in most executive processing that occurs in the brain. Theta burst stimulation (TBS) is a paradigm of TMS which has been shown to effectively modulate WM. Moreover, TBS can modulate gamma neural oscillations in the brain and neural activity, both of which have been implicated in the physiology of WM and pathophysiology of the disease process in schizophrenia, making these measures highly valuable for assessing physiological effects of TBS on cognition, quality of life and cortical inhibition. The purpose of this study is to evaluate the effect of TBS on WM in patients with schizophrenia, to develop evidence for potential brain stimulation techniques to treat cognitive deficits in schizophrenia.

Study activities and population group: Study subjects will be inpatient schizophrenic individuals with minimal positive symptoms and predominant cognitive deficits at Duke University Hospital. In an initial session they will be screened and taught a WM task. Following this, one TBS session will follow in which TBS will target dorsolateral prefrontal cortex. They will perform the WM task before, with and after the TBS, with an expected pre-post enhancement of WM performance.

Implications - There is a great need for treatments for cognitive deficits in schizophrenia. The results of this study will serve to generate pilot data for a much larger grant to develop a TBS therapy for remediating such cognitive deficits.

DETAILED DESCRIPTION:
Purpose of the study Aim1: Evaluate the effect of theta burst stimulation (TBS) on working memory (WM) in patients with schizophrenia. Hypothesis 1 - There will be significant improvement in WM compared to baseline with one session of TBS.

Background and Significance Schizophrenia is an illness known to have cognitive deficits, with a chronic and variable course. There is extensive research on cognitive deficits, with working memory, processing speed and verbal memory being some of the domains affected. Some modalities of treatment that have been tried to reverse these cognitive deficits are medications and cognitive behavioral therapy with minimal benefits. A few studies have shown modulation of working memory with routine repetitive transcranial magnetic stimulation at frequencies not exceeding 10 to 20 Hz of stimulation. Other studies have shown the working memory to be related to gamma oscillations. A few studies have also shown that transcranial magnetic stimulation (TMS) modulates these gamma oscillations as well. There is an extensive body of literature that shows that working memory has contributions from theta and gamma oscillations in the brain. Theta burst stimulation (TBS) is a form of transcranial magnetic stimulation (TMS), that entrains gamma and theta frequencies in the brain. It could be the most appropriate form of brain stimulation for improving cognition in schizophrenia patients because it has been shown to modulate brain oscillations in small samples of patients. The area for targeting would be the dorsolateral prefrontal cortex which is the site of origin of the gamma oscillations and plays a significant role in working memory.

Design and Procedures The study is designed to be a pilot one evaluating the effect of TBS on WM in patients with schizophrenia. The investigators plan to screen 20 subjects to have 10 participants. Working memory will be tested using delayed match sample task (DMS) and brief assessment of cognition in schizophrenia battery (BACS).

Transcranial Magnetic Stimulation (TMS) administration The patient would be transported from the inpatient unit to the TMS lab following screening and consent process. They would be accompanied by nursing staff. During their visit to the TMS lab a sample TMS session including motor threshold determination will be conducted. Subjects would be allowed to practice the DMS task to allow for the ceiling in practice effect of the task. The BACS would be administered before and after the TMS session.

Treatment Sessions Subjects would be administered left sided theta burst stimulation (TBS).The subject will be seated in a chair. A 64-channel electrode cap may be applied to the head for EEG recording. Electromyogram (EMG) electrodes will be applied to the right hand for motor evoked potential (MEP) recording. Subjects will perform the DMS task while sitting in the chair during the TMS session. EEG and EMG will be recorded throughout the treatment sessions. For theta burst stimulation the active motor threshold would be 80 % as used in most theta burst studies detailed in this review. Subjects would receive theta burst stimulation comprising 50 Hz bursts given at 3 to 5 Hz for close to 10 minutes which comprises 60 trains and 1800 pulses. The subject will be monitored until MEPs return to baseline. A side effects checklist will be completed at the beginning and at the end of the experimental session. All sessions will be performed by one of the protocol investigators, or by a trained and accredited research assistant supervised by the protocol investigators.

Clinical and cognitive assessments/tasks PANSS The Positive and negative symptoms scale is used to assess the severity of schizophrenia. It has three subscales - positive, negative and general psychopathology. Each of these subscales had 7 items, the maximum scores on each of these subscales in 49, minimum score being 7.

DMS task The DMS task is a modified version of the Sternberg task and has been adapted for use in cognitive paradigms accompanying transcranial magnetic stimulation. Each trial will last 13 s, with the following sequence of three task stages: encoding, retention and probe stages.

BACS - Tasks to be done from the actual BACS battery of tests List Learning (Verbal Memory). Patients are presented with 15 words and then asked to recall as many as possible. This procedure is repeated 5 times. There are two alternate forms.

Digit Sequencing Task (verbal working Memory). Patients are presented with clusters of numbers of increasing length. They are asked to tell the experimenter the numbers in order, from lowest to highest.

Token Motor Task (Motor Speed). Patients are given 100 plastic tokens and asked to place them into a container as quickly as possible for 60 seconds.

Verbal Fluency. Tests of Category Instances (Semantic Fluency) and Controlled Oral Word Association Test (Letter Fluency) are administered. Patients are given 60 seconds to name as many words as possible within a given semantic category, and in two separate trials, patients are given 60 seconds to generate as many words as possible that begin with a given letter. The total number of words from the three trials is the outcome measure.

Tower of London (Reasoning and Problem Solving). Patients look at two pictures simultaneously. Each picture shows 3 different-colored balls arranged on 3 pegs, with the balls in a unique arrangement in each picture. The patients are told about the rules in the task and are asked to provide the least number of times the balls in one picture would have to be moved to make the arrangement of balls identical to that of the other, opposing picture. There are two alternate forms.

Symbol Coding (Attention and Processing Speed). As quickly as possible, patients write numerals 1-9 as matches to symbols on a response sheet for 90 seconds.

Each of the six measures are compared to a healthy control sample to create z-scores, and a composite score is calculated by summing these z-scores and calculating a z-score of that sum. The composite score has high test-retest reliability in patients with schizophrenia and healthy controls (ICCs > .80).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years of age with schizophrenia or schizoaffective disorder
* No other mental health diagnoses
* Right handed males and females
* May have mild positive symptoms (score of </= 21)
* May have negative symptoms
* Ability to provide informed consent
* No restriction on concomitant medications given

Exclusion Criteria:

* Intellectual disability
* Any organic brain illness Presence of dementia symptoms or traumatic brain injury Primary diagnosis of substance use Seizure disorder Actively symptomatic with PANSS positive symptom sub-scale >21. Concurrently receiving electroconvulsive therapy (ECT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green MF, Nuechterlein KH, Gold JM, Barch DM, Cohen J, Essock S, Fenton WS, Frese F, Goldberg TE, Heaton RK, Keefe RS, Kern RS, Kraemer H, Stover E, Weinberger DR, Zalcman S, Marder SR. Approaching a consensus cognitive battery for clinical trials in schizophrenia: the NIMH-MATRICS conference to select cognitive domains and test criteria. Biol Psychiatry. 2004 Sep 1;56(5):301-7. doi: 10.1016/j.biopsych.2004.06.023. PMID 15336511
- [Background] Keefe RS, Fox KH, Harvey PD, Cucchiaro J, Siu C, Loebel A. Characteristics of the MATRICS Consensus Cognitive Battery in a 29-site antipsychotic schizophrenia clinical trial. Schizophr Res. 2011 Feb;125(2-3):161-8. doi: 10.1016/j.schres.2010.09.015. Epub 2010 Dec 31. PMID 21075600
- [Background] Young JW, Geyer MA. Developing treatments for cognitive deficits in schizophrenia: the challenge of translation. J Psychopharmacol. 2015 Feb;29(2):178-96. doi: 10.1177/0269881114555252. Epub 2014 Dec 16. PMID 25516372
- [Background] Barr MS, Farzan F, Arenovich T, Chen R, Fitzgerald PB, Daskalakis ZJ. The effect of repetitive transcranial magnetic stimulation on gamma oscillatory activity in schizophrenia. PLoS One. 2011;6(7):e22627. doi: 10.1371/journal.pone.0022627. Epub 2011 Jul 27. PMID 21818354
- [Background] Farzan F, Barr MS, Sun Y, Fitzgerald PB, Daskalakis ZJ. Transcranial magnetic stimulation on the modulation of gamma oscillations in schizophrenia. Ann N Y Acad Sci. 2012 Aug;1265:25-35. doi: 10.1111/j.1749-6632.2012.06543.x. Epub 2012 Jul 23. PMID 22823464
- [Background] Hasan A, Brinkmann C, Strube W, Palm U, Malchow B, Rothwell JC, Falkai P, Wobrock T. Investigations of motor-cortex cortical plasticity following facilitatory and inhibitory transcranial theta-burst stimulation in schizophrenia: a proof-of-concept study. J Psychiatr Res. 2015 Feb;61:196-204. doi: 10.1016/j.jpsychires.2014.12.006. Epub 2014 Dec 19. PMID 25555304
- [Background] Tikka SK, Nizamie SH, Venkatesh Babu GM, Aggarwal N, Das AK, Goyal N. Safety and Efficacy of Adjunctive Theta Burst Repetitive Transcranial Magnetic Stimulation to Right Inferior Parietal Lobule in Schizophrenia Patients With First-Rank Symptoms: A Pilot, Exploratory Study. J ECT. 2017 Mar;33(1):43-51. doi: 10.1097/YCT.0000000000000343. PMID 27428476
- [Background] Demirtas-Tatlidede A, Freitas C, Cromer JR, Safar L, Ongur D, Stone WS, Seidman LJ, Schmahmann JD, Pascual-Leone A. Safety and proof of principle study of cerebellar vermal theta burst stimulation in refractory schizophrenia. Schizophr Res. 2010 Dec;124(1-3):91-100. doi: 10.1016/j.schres.2010.08.015. PMID 20817483
- [Background] Gonzalez-Burgos G, Cho RY, Lewis DA. Alterations in cortical network oscillations and parvalbumin neurons in schizophrenia. Biol Psychiatry. 2015 Jun 15;77(12):1031-40. doi: 10.1016/j.biopsych.2015.03.010. Epub 2015 Mar 17. PMID 25863358
- [Background] Barr MS, Farzan F, Rusjan PM, Chen R, Fitzgerald PB, Daskalakis ZJ. Potentiation of gamma oscillatory activity through repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex. Neuropsychopharmacology. 2009 Oct;34(11):2359-67. doi: 10.1038/npp.2009.79. Epub 2009 Jul 15. PMID 19606086
- [Background] Keefe RS, Poe M, Walker TM, Harvey PD. The relationship of the Brief Assessment of Cognition in Schizophrenia (BACS) to functional capacity and real-world functional outcome. J Clin Exp Neuropsychol. 2006 Feb;28(2):260-9. doi: 10.1080/13803390500360539. PMID 16484097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 6 patients with diagnoses of schizophrenia, which included 4 inpatients and 2 outpatients.
Groups:
- Patients With a Diagnosis of Schizophrenia: We recruited 6 patients with diagnoses of schizophrenia. Inpatient subjects were recruited towards the latter half of their inpatient stay, after their positive symptoms had decreased in severity. PANSS was performed at recruitment and subjects were chosen for the study only if their positive symptom score was less than or equal to 21. Our other inclusion criteria for the study were patients in the age group of 18-50 years, right handed, with no other comorbid DSM-5 diagnoses (including substance use disorder), and able to give informed consent. Subjects with organic basis for their psychopathology or intellectual disability, were excluded from the study.
  Intervention administered - Theta Burst Stimulation (TBS) with Brief Assessment of Cognition in Schizophrenia (BACS) administered before and after TBS.
Period: Overall Study
Arm/Group | Patients With a Diagnosis of Schizophrenia
Started | 6
Completed | 3
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- Patients With a Diagnosis of Schizophrenia: We recruited 6 patients with diagnoses of schizophrenia. Inpatient subjects were recruited towards the latter half of their inpatient stay, after their positive symptoms had decreased in severity. PANSS was performed at recruitment and subjects were chosen for the study only if their positive symptom score was less than or equal to 21. Our other inclusion criteria for the study were patients in the age group of 18-50 years, right handed, with no other comorbid DSM-5 diagnoses (including substance use disorder), and able to give informed consent. Subjects with organic basis for their psychopathology or intellectual disability, were excluded from the study.
Arm/Group | Patients With a Diagnosis of Schizophrenia
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Brief Assessment of Cognition (BACS) Composite T Score [Mean (Standard Deviation); unit: Composite T- Score] | 26.3 (17.4)

OUTCOME MEASURES:

1. Primary Outcome: Brief Assessment of Cognition (BACS) Composite T Score
Description: Performance on tasks included in the Brief Assessment of Cognition in Schizophrenia (BACS) battery, task performed and results recorded on IPAD. The mean change from baseline in total cognitive score on the BACS was calculated as a weighted average of T-scores (normalized for age) from BACS subtests including Verbal Memory, Digit Sequencing, Token Motor, Symbol Coding, Semantic Fluency, Letter Fluency, and Tower of London. The minimum and maximum values possible for this composite T-score of the change from baseline were -131 and 131, respectively. Higher values (positive changes from baseline) indicate better performance.
Time Frame: 30 minutes
Measure: Mean (95% Confidence Interval); unit: Composite T- Score
Arm/Group | Theta Burst Stimulation Arm
Number analyzed (Participants) | 3
Composite T- Score | 37.33 [18.5 to 56.1]

2. Secondary Outcome: Change in Gamma and Theta Oscillations as Measured by EEG
Time Frame: one session, approximately 30 minutes
Population: No EEG data was collected
Arm/Group | Theta Burst Stimulation Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With a Diagnosis of Schizophrenia
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT03288779/Prot_SAP_000.pdf